CLINICAL TRIAL: NCT03290742
Title: Incidence of and Risk Factors for Perioperative Infection Among Patients Undergoing Radical Cystectomy
Brief Title: Infection Among Patients Undergoing Radical Cystectomy.
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Krystian Kaczmarek, Principal Investigator, Pomeranian Medical University Szczecin
Other Study IDs: INF1
Record Dates: First submitted 2017-09-14; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Cystostomy Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without documented infection.: Patients without infection during 30 day follow-up after radical cystectomy.
- Patients with documented infection.: Patients with documented any kind of infection (urinary tract infection, blood infection/septic shock, surgical site infection) during 30 day follow-up after radical cystectomy.

SUMMARY:
Investigators plan to perform a review of medical records a single urology department to identify patients with febrile perioperative infection who underwent radical cystectomy and urinary diversion for bladder cancer from January 2014 to July 2017.

Investigators plan assess a potential variables to find correlation with infections after surgery.

Characteristics, including age, sex, length of hospital stay, body mass index (BMI), diabetes, hypertension, estimated glomerular filtration rate (eGFR), preoperative hydronephrosis, smoking status, neoadjuvant chemotherapy, pathological stage, lymph node involvement, types of urinary diversion, operative method (open/laparoscopic), operative time and receipt of a perioperative blood transfusion (PBT) will be asses as potential risk factor for perioperative infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent radical cystectomy and urinary diversion for bladder cancer.

Exclusion Criteria:

* documented infection at the time of radical cystectomy
* concurrent organ resection such as nephrectomy, nephroureterectomy
* partial cystectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent radical cystectomy and urinary diversion for bladder cancer from January 2014 to July 2017.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2017-08-20 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with perioperative infection after radical cystectomy. | 30 days
  A review of medical records in a single urology department will be performed to identified all participants with perioperative infection after radical cystectomy.

SECONDARY OUTCOMES:
Association between perioperative infection after radical cystectomy and patients' age. | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and sex. | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and length of hospital stay. | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and body mass index. | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and diabetes. | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and hypertension. | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and estimated glomerular filtration rate | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and preoperative hydronephrosis. | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and smoking status. | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and neoadjuvant chemotherapy. | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and pathological stage. | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and lymph node involvement. | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and types of urinary diversion. | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and operative method (open/laparoscopic). | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and operative time. | 30 days
  Logistic regression analysis.
Association between perioperative infection after radical cystectomy and receipt of a perioperative blood transfusion. | 30 days
  Logistic regression analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology and Urological Oncology, Szczecin, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No